CLINICAL TRIAL: NCT05596279
Title: Clinical Performance of a Novel Hybrid Intravascular Ultrasound-Optical Coherence Tomography System: a Prospective Randomized Controlled Clinical Trial
Brief Title: PANOVISION: Feasibility and Safety of Hybrid IVUS-OCT System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harbin Medical University (Other)
Collaborators: Second Hospital of Jilin University (Other); Wuhan Asia Heart Hospital (Other); Panorama Hengsheng (Beijing) Science and Technology Co., Ltd. (Unknown)
Responsible Party: Principal Investigator, Yu Bo, Director of Department of Cardiology, The Second Affiliated Hospital of Harbin Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: VP-3003-1901
Record Dates: First submitted 2022-10-20; First posted 2022-10-27 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Coronary Artery Disease; Intravascular Imaging Device
Keywords: Hybrid imaging; Intravascular ultrasound; Optical coherence tomography
MeSH Terms: conditions — Coronary Artery Disease | interventions — Ultrasonography, Interventional; Tomography, Optical Coherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravascular ultrasound (Experimental): Hybrid IVUS-OCT and control IVUS were performed after stenting
  Interventions: Diagnostic Test: Intravascular ultrasound
- Optical coherence tomography (Experimental): Hybrid IVUS-OCT and control OCT were performed after stenting
  Interventions: Diagnostic Test: Optical coherence tomography

INTERVENTIONS:
Diagnostic Test: Intravascular ultrasound — Hybrid IVUS-OCT and control IVUS were performed after stenting
  Arms: Intravascular ultrasound
Diagnostic Test: Optical coherence tomography — Hybrid IVUS-OCT and control OCT were performed after stenting
  Arms: Optical coherence tomography

SUMMARY:
Intravascular ultrasound (IVUS) and optical coherence tomography (OCT) were all recommended for percutaneous coronary intervention (PCI) optimization in the latest guidelines, however, which imaging modality was more suitable as either a diagnostic or guidance tool was still unknown. Recently, a novel, well-designed hybrid imaging system was approved for clinical use, allowing the accurate co-registration of two imaging modalities and immediate, simultaneous image review. For testing each modality in the hybrid imaging system, the investigators conducted this prospective, multicentre, non-inferiority trial. In this study, all participants achieved hybrid IVUS-OCT imaging after stenting, at meanwhile, patients randomly assigned to the IVUS arm were performed control IVUS (OptiCross, Boston Scientific, Natick, MA), and patients randomly assigned to the OCT arm were performed control OCT (C7 Dragonfly Duo, St. Jude Medical, St. Paul, MN). In this study, the investigators evaluated the non-inferiority of standalone IVUS versus control IVUS or standalone OCT versus control OCT in clinical feasibility using clear stent capture rate (CSCR) and safety using perioperative device-related adverse cardiovascular events.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years
* Patients eligible for elective percutaneous coronary intervention
* Understand and voluntarily sign the informed consent form

Exclusion Criteria:

The lesion-related exclusion criteria:

* More than 1 stent was planned to deploy in culprit lesion
* In-stent restenosis
* Bifurcation lesion with proposed double stent implantation
* The length of the reference vessel segment proximal or distal to the lesion was less than 5mm
* The length of the implanted stent was larger than 33mm
* The diameter of reference vessel was less than 2 mm or larger than 4 mm
* Lesions were in left main or ostium of right coronary artery
* The distance between either end of the lesion and the lateral branches larger than 2 mm in diameter was less than 5 mm
* Angiography revealed thrombosis in culprit vessel
* Severely calcified lesions or tortuous coronary arteries
* Decreased blood flow (thrombolysis in myocardial infarction score ≤ 2)

Patients-level exclusion criteria:

* Breastfeeding or pregnant women, the subject (or his partner) who had a pregnancy plan during the trial or within 6 months after the end of the trial, and subject who did not agree to use contraception during the trial
* Participants who had withdrawn from other clinical studies within 3 months or are participating in other clinical trials
* Acute myocardial infarction occurred within one week prior to screening
* Cardiac troponin I or cardiac troponin T levels exceed the upper limit of normal reference values within 72 hours of procedure and were of clinical significance
* Renal insufficiency with creatinine > 200μmol/L
* Unsuitable for coronary artery bypass grafting (CABG)
* Unsuitable for percutaneous coronary intervention;
* Coronary spasm
* Chronic total occlusion or subtotal occlusion
* Severe hemodynamic disturbances or shock
* History of CABG
* Coagulation is abnormal and clinically significant
* Severe heart failure (NYHA III, IV or Left ventricular ejection fraction < 30%)
* History of contrast allergy
* Multi-vessel disease
* Chemotherapy or planned chemotherapy
* Investigators consider unsuitable for participants selected for this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-11-20 (Actual); Primary Completion 2020-08-12 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Clear stent capture rate (CSCR) | During the procedure
  The CSCR detected was defined as the ratio of the clear stent length to the total stent length

SECONDARY OUTCOMES:
Proportion of patients with clear image length ≥ 24mm | During the procedure
  Measured by IVUS, OCT and hybrid IVUS-OCT
Detection rate of edge dissection, tissue prolapse and stent malapposition | During the procedure
  Assessed by IVUS, OCT and hybrid IVUS-OCT
Device success rate | During the procedure
  Device success is defined as well-manipulated and capable of acquiring intravascular images
Adverse procedure-related adverse cardiovascular events | Periprocedure
  Coronary spasm, acute vessel occlusion, coronary dissection, or thrombosis

CONTACTS AND LOCATIONS:
Overall Officials: Bo Yu, MD, PhD, Study Chair — The Second Affiliated Hospital of Harbin Medical University; Bin Liu, MD, PhD, Principal Investigator — Second Hospital of Jilin University; Xi Su, MD, PhD, Principal Investigator — Wuhan Asia Heart Hospital
Locations (3):
- China (3):
  - The Second Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Wuhan Asia Heart Hospital, Wuhan, Hubei
  - The Second Hospital of Jilin University, Changchun, Jilin

IPD SHARING:
Plan to Share IPD: No